CLINICAL TRIAL: NCT01887366
Title: A 12-week, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Once-Weekly Intra-Muscular Injections of TV-1380 (150 mg/Week or 300 mg/Week) as Treatment for Facilitation of Abstinence in Cocaine-Dependent Subjects
Brief Title: Efficacy and Safety of TV-1380 as Treatment for Facilitation of Abstinence in Cocaine-Dependent Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TV1380-COA-201
Record Dates: First submitted 2013-06-24; First posted 2013-06-26 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-10

CONDITIONS: Cocaine Addiction
Keywords: Cocaine addiction; TV-1380; Recombinant human serum albumin (HSA) mutated butyrylcholinesterase (AlbuBChE)
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — TV-1380

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- TV-1380 150 mg (Experimental)
  Interventions: Drug: TV-1380 150 mg
- TV-1380 300 mg (Experimental)
  Interventions: Drug: TV-1380 300 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TV-1380 150 mg — Subjects assigned to TV-1380 150 mg will be administered one intra-muscular (IM) injection once weekly over 12 weeks. The injection volume will be the same for all treatment groups. Therefore, to accommodate the volume required for the highest dosing group (3.0 mL), subjects in this group will receive 3.0 mL IM injection of TV-1380 150 mg (1.5 mL TV-1380 and 1.5 mL placebo/diluents).
  Other Names: Recombinant human serum albumin (HSA) mutated butyrylcholinesterase (AlbuBChE)
  Arms: TV-1380 150 mg
Drug: TV-1380 300 mg — Subjects assigned to TV-1380 300 mg will be administered one intra-muscular (IM) injection once weekly over 12 weeks. Subjects in this treatment group will receive 3.0 mL TV-1380.
  Other Names: Recombinant human serum albumin (HSA) mutated butyrylcholinesterase (AlbuBChE)
  Arms: TV-1380 300 mg
Drug: Placebo — Subjects assigned to placebo will be administered one intra-muscular (IM) injection once weekly over 12 weeks. Subjects in this treatment group will receive 3.0 mL placebo.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to assess the efficacy and safety of TV-1380 [Recombinant human serum albumin (HSA) mutated butyrylcholinesterase (AlbuBChE)] in facilitating abstinence in cocaine-dependent subjects.

ELIGIBILITY:
Inclusion Criteria:

* Have the ability to understand, and having understood, provide written informed consent to comply with the treatment protocol.
* Male or female aged 18-60 years (inclusive).
* Meet Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition.
* Other criteria apply; please contact the site for more information.

Exclusion Criteria:

* Meet criteria for current dependence on any psychoactive substance other than cocaine, alcohol, nicotine, benzodiazepines, or marijuana OR have physiological dependence on alcohol requiring detoxification.
* Are currently treated with an opiate-substitute (buprenorphine or methadone) maintenance treatment or received therapy with any opiate-substitute within 90 days preceding screening.
* Have one or more severe psychiatric disorders as determined by the Mini International Neuropsychiatric Interview (MINI) such as psychosis, schizophrenia, bipolar disease, major depression, or eating disorders in screening.
* Have one or more major neurologic disorders such as dementia or organic brain disease.
* Have other serious medical illnesses (including but not limited to uncontrolled hypertension, significant heart disease, respiratory disease including asthma, hepatic disease, renal disease, AIDS) or other potentially life threatening or progressive medical illness that may compromise subject safety or study conduct as determined by the site MD.
* Other criteria apply; please contact the site for more information.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 208 (Actual)
Dates: Start 2013-06; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Urine test for cocaine | Treatment Phase weeks 10 - 12

SECONDARY OUTCOMES:
Percent of urine samples that are considered negative for cocaine metabolites. | Treatment Phase Weeks 5 -12
Summary of participants with adverse events | From signing of the informed consent form to the end of the follow-up period (Week 16)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (14):
  - Teva Investigational Site 10663, Los Angeles, California
  - Teva Investigational Site 10665, Oceanside, California
  - Teva Investigational Site 10659, San Francisco, California
  - Teva Investigational Site 10746, Torrance, California
  - Teva Investigational Site 10664, North Miami, Florida
  - Teva Investigational Site 10661, Boston, Massachusetts
  - Teva Investigational Site 10668, New Bedford, Massachusetts
  - Teva Investigational Site 10747, St Louis, Missouri
  - Teva Investigational Site 10745, Las Vagas, Nevada
  - Teva Investigational Site 10667, Marlton, New Jersey
  - Teva Investigational Site 10662, Columbus, Ohio
  - Teva Investigational Site 10660, Pittsburgh, Pennsylvania
  - Teva Investigational Site 10658, Charleston, South Carolina
  - Teva Investigational Site 10666, Salt Lake City, Utah
- Spain (5):
  - Teva Investigational Site 31064, Alicante
  - Teva Investigational Site 31063, Barcelona
  - Teva Investigational Site 31065, Barcelona
  - Teva Investigational Site 31069, Barcelona
  - Teva Investigational Site 31068, Madrid